CLINICAL TRIAL: NCT04387773
Title: Effect of GOCOVRI on Quantity and Quality of Gait in Parkinson's Disease
Brief Title: Effect of GOCOVRI (Amantadine, Extended Release Capsules) on Gait in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Adamas Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Amie Hiller, MD, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20105
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Amantadine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GOCOVRI Treatment (Experimental): All participants will have gait, balance, dyskinesia assessed before and after receiving GOCOVRI (274 mg/day).
  Interventions: Drug: GOCOVRI

INTERVENTIONS:
Drug: GOCOVRI — Participants will have gait and balance baseline assessment and then repeat assessment after being on full-dose of GOCOVRI for two weeks. The assessments will include measures of gait, balance and dyskinesia. Participants will also wear body-worn sensors (on wrist, feet and lumbar area) during daily-life for seven days to quantify mobility.
  GOCOVRI will be started at 137mg/day for two weeks and then increased to 274mg/day for two weeks. Participants will repeat baseline assessments and then decrease to a dose of 137mg/day of GOCOVRI for one week, before stopping the medication completely.
  All participants will receive GOCOVRI and they will know that they are on study drug. No placebo group.

SUMMARY:
The purpose of the study is to learn about the effect of GOCOVRI (Amantadine extended release) on activity levels and measures of gait and balance quality in people with Parkinson's disease (PD) and levodopa induced dyskinesia (LID) during daily activities using body-worn sensors.

DETAILED DESCRIPTION:
Levodopa induced dyskinesia (LID) is a symptom of Parkinson's disease for which there are limited treatment options. LID leads to reduced quality of life, increased caregiver burden and an increased risk of falls (Rascol et al., 2015, Chapuis et al., 2005). GOCOVRI™ is an extended release capsule prescription medication shown to reduce LID in people with PD (Pahwa et al., 2017, Pahwa et al., 2018). However, a number of studies have identified an increase in falls in those on the active medication study arm but not the placebo arm (13% increase in active and 7% in placebo) (Pahwa et al., 2017). In order to understand this increase in falls, comprehensive measurements of quantity of activity (gait measured in the home environment) and quality of activity (comprehensive gait characteristics that may increase risk of falls) need to be assessed in participants taking GOCOVRI™. In addition, the evidence for the effect of GOCOVRI™ on gait and balance in PD is limited (Smulders et al., 2016).

This study is an open label study in which the following Aims will be studied:

Aim I: Investigate the effect of GOCOVRI™ on activity levels in people with Parkinson's disease (PD) and Levodopa induced dyskinesia (LID) Hypothesis I: We hypothesize that GOCOVRI™ will result in an increase of daily activity due to improvement in LID symptoms. Primary outcome measures: Total amount of activity per day

Aim II: Investigate the effect of GOCOVRI™ on comprehensive measures of gait and balance quality in people with PD with LID Hypothesis II: We hypothesize GOCOVRI™ may improve discrete characteristics of gait and balance that is evident even within the first hour of the day walking.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson'd Disease in accordance with the United Kingdom (UK) Brain Bank Criteria
* Hoehn & Yahr scores of II-IV
* subjective report of experiencing at least 1hr/day (two, half-hour periods) of ON time with troublesome Levodopa-Induced Dyskinesia (LID)
* ambulation with or without aids (e.g., walker or cane)
* ≥30 days of a stable regimen of anti-Parkinson's medications that includes a levodopa dose administered ≥3 times daily
* a stable dose of levodopa throughout the study
* no amantadine for a minimum of 30 days prior to enrollment in the study

Exclusion Criteria:

* neurological or musculoskeletal disorders
* orthostatic hypotension at screening (defined as a drop of ≥20mm mercury (HG) systolic and ≥10mm HG diastolic at 2 or 5 minutes of quiet standing after 5 minutes of supine rest)
* a major psychotic disorder
* contraindication to GOCOVRI™ at time of screening, especially renal impairment estimated by glomerular filtration rate (eGFR) < 50 ml/min/1.73 m2) as impaired renal function can increase the chances of adverse reactions to the study drug
* mild to severe cognitive impairment as measured by Montreal Cognitive Assessment (MoCA) score ≤ 23
* concurrent use of immediate release amantadine
* are pregnant or plan to become pregnant
* an implanted deep brain stimulator

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amie Hiller, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participants' data will be available (including data dictionary) after de-identification and will include all data collected during the trial. The study protocol, statistical analysis plan, informed consent, clinical study report, and analytic code will all be available 3 months after study publication to 5 years after publication. This data will be shared with anyone providing a methodologically sound proposal. To gain access to the data proposals should be directed to carlsonp@ohsu.edu and requesters will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 3 months to 5 years after study publication
Access Criteria: Requesters will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Groups:
- GOCOVRI Treatment: All participants will have gait, balance, dyskinesia assessed before and after receiving GOCOVRI (274 mg/day).
  GOCOVRI: Participants will have gait and balance baseline assessment and then repeat assessment after being on full-dose of GOCOVRI for two weeks. The assessments will include measures of gait, balance and dyskinesia. Participants will also wear body-worn sensors (on wrist, feet and lumbar area) during daily-life for seven days to quantify mobility.
  GOCOVRI will be started at 137mg/day for two weeks and then increased to 274mg/day for two weeks. Participants will repeat baseline assessments and then decrease to a dose of 137mg/day of GOCOVRI for one week, before stopping the medication completely.
  All participants will receive GOCOVRI and they will know that they are on study drug. No placebo group.
Period: Overall Study
Arm/Group | GOCOVRI Treatment
Started | 8
Completed | 5
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | GOCOVRI Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 7
Age, Continuous [Mean (Full Range); unit: years] | 70.9 [60 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
Years since Parkinson's disease diagnosis [Mean (Full Range); unit: years] | 9.25 [5 to 15]
Years with levodopa induced dyskinesias [Mean (Full Range); unit: years] | 3 [0 to 4]
Participants with one or more falls in the last 12-months [Count of Participants; unit: Participants] | 6

OUTCOME MEASURES:

1. Primary Outcome: Aim I: Investigate the Effect of GOCOVRI™ on Activity Levels in People With Parkinson's Disease (PD) and Levodopa Induced Dyskinesia (LID) Measure: Number of Walking Bouts Per Hour
Description: Aim I: Investigate the effect of GOCOVRI™ on activity levels in people with Parkinson's disease (PD) and Levodopa induced dyskinesia (LID).
  Hypothesis I: We hypothesized that GOCOVRI™ would result in an increase of daily activity due to improvement in LID symptoms.
  Measure: number of walking bouts per hour
Time Frame: Baseline and on drug; one week of daily life monitoring at each time point
Population: 1 participant that completed the protocol was not included for analysis due to incomplete data
Measure: Mean (Standard Deviation); unit: Average number of walking bouts per hour
Arm/Group | GOCOVRI Treatment
Number analyzed (Participants) | 4
Average number of walking bouts per hour
  Baseline | 9.98 (6.23)
  On drug | 7.68 (4.86)
Statistical Analysis 1: Comparison: GOCOVRI Treatment; We hypothesized that GOCOVRI would result in an increase of daily activity due to improvement in LID symptoms; Test type: Superiority; p > .05, t-test, 2 sided; Mean Difference (Final Values) = 2.3

2. Primary Outcome: Aim I: Investigate the Effect of GOCOVRI™ on Activity Levels in People With Parkinson's Disease (PD) and Levodopa Induced Dyskinesia (LID) Measure: Number of Turns Per Hour
Description: Aim I: Investigate the effect of GOCOVRI™ on activity levels in people with Parkinson's disease (PD) and Levodopa induced dyskinesia (LID).
  Hypothesis I: We hypothesized that GOCOVRI™ would result in an increase of daily activity due to improvement in LID symptoms.
  Measure: number of turns per hour
Time Frame: Baseline and on drug; one week of daily life monitoring at each time point
Population: 1 participant that completed the protocol was not included for analysis due to incomplete data
Measure: Mean (Standard Deviation); unit: Average number of turns per hour
Arm/Group | GOCOVRI Treatment
Number analyzed (Participants) | 4
Average number of turns per hour
  Baseline | 84.78 (18.47)
  On drug | 69.8 (31.92)
Statistical Analysis 1: Comparison: GOCOVRI Treatment; We hypothesized that GOCOVRI would result in an increase of daily activity due to improvement in LID symptoms; Test type: Superiority; p > .05, t-test, 2 sided; Mean Difference (Final Values) = 14.98

3. Primary Outcome: Aim I: Investigate the Effect of GOCOVRI™ on Activity Levels in People With Parkinson's Disease (PD) and Levodopa Induced Dyskinesia (LID) Measure: Total Number of Turns During the Day
Description: Aim I: Investigate the effect of GOCOVRI™ on activity levels in people with Parkinson's disease (PD) and Levodopa induced dyskinesia (LID).
  Hypothesis I: We hypothesized that GOCOVRI™ would result in an increase of daily activity due to improvement in LID symptoms.
  Measure: total number of turns during the day
Time Frame: Baseline and on drug; one week of daily life monitoring at each time point
Population: 1 participant that completed the protocol was not included for analysis due to incomplete data
Measure: Mean (Standard Deviation); unit: Total number of turns per day
Arm/Group | GOCOVRI Treatment
Number analyzed (Participants) | 4
Total number of turns per day
  Baseline | 6540.7 (3024.5)
  On drug | 4147.5 (2188.9)
Statistical Analysis 1: Comparison: GOCOVRI Treatment; Test type: Superiority; p = 0.037, t-test, 2 sided; Mean Difference (Final Values) = 2393.2

4. Primary Outcome: Aim II: Investigate the Effect of GOCOVRI™ on Comprehensive Measures of Gait and Balance Quality in People With PD With LID Measure: Variability in the Turn Rate Per Step (CoV, Coefficient of Variation)
Description: Aim II: Investigate the effect of GOCOVRI™ on comprehensive measures of gait and balance quality in people with PD with LID Hypothesis II: We hypothesize GOCOVRI™ may improve discrete characteristics of gait and balance that is evident even within the first hour of the day walking.
  Measure: Variability in the turn rate per step (CoV, Coefficient of Variation) Collection methods: wearable sensors worn during daily life used to measure participant walking characteristics; analysis extracts bouts of walking and turning, and specific gait measures for each are averaged across the weeklong collections; CoV calculated using standard deviation and mean of turn rate per step
Time Frame: Baseline and on drug; one week of daily life monitoring at each time point
Population: 1 participant that completed the protocol was not included for analysis due to incomplete data
Measure: Median (Full Range); unit: CoV, unitless (mean divided by Standard)
Arm/Group | GOCOVRI Treatment
Number analyzed (Participants) | 4
CoV, unitless (mean divided by Standard)
  Baseline | 0.39 [0.37 to 0.43]
  On drug | 0.42 [0.38 to 0.45]
Statistical Analysis 1: Comparison: GOCOVRI Treatment; Test type: Superiority; p = 0.012, t-test, 2 sided; Mean Difference (Final Values) = 0.03

5. Primary Outcome: Aim II: Investigate the Effect of GOCOVRI™ on Comprehensive Measures of Gait and Balance Quality in People With PD With LID Measure: Variability in Total Number of Steps During Turns (CoV, Coefficient of Variation)
Description: Aim II: Investigate the effect of GOCOVRI™ on comprehensive measures of gait and balance quality in people with PD with LID Hypothesis II: We hypothesize GOCOVRI™ may improve discrete characteristics of gait and balance that is evident even within the first hour of the day walking.
  Measure: variability in total number of steps during turns (CoV, Coefficient of Variation) Collection methods: wearable sensors worn during daily life used to measure participant walking characteristics; analysis extracts bouts of walking and turning, and specific gait measures for each are averaged across the weeklong collections; CoV calculated using standard deviation and mean of the number of steps to complete turns
Time Frame: Baseline and on drug; one week of daily life monitoring at each time point
Population: 1 participant that completed the protocol was not included for analysis due to incomplete data
Measure: Median (Full Range); unit: CoV, unitless (mean divided by Standard)
Arm/Group | GOCOVRI Treatment
Number analyzed (Participants) | 4
CoV, unitless (mean divided by Standard)
  Baseline | 0.55 [0.50 to 0.67]
  On drug | 0.53 [0.48 to 0.63]
Statistical Analysis 1: Comparison: GOCOVRI Treatment; Test type: Superiority; p = 0.047, t-test, 2 sided; Mean Difference (Final Values) = 0.02

ADVERSE EVENTS:
Time Frame: Adverse events were followed for the 6-weeks of study participation.
Description: Definitions did not differ
Groups:
- GOCOVRI Half Dose (Week 0-2); GOCOVRI Full Dose (Week 2-4); GOCOVRI Half Dose (Week 4-5): Participants will have gait and balance baseline assessment and then repeat assessment after being on full-dose of GOCOVRI for two weeks. The assessments will include measures of gait, balance and dyskinesia. Participants will also wear body-worn sensors (on wrist, feet and lumbar area) during daily-life for seven days to quantify mobility.
  GOCOVRI will be started at 137mg/day for two weeks (half dose) and, if tolerated, increased to 274mg/day for two weeks (full dose). Participants will repeat assessments and then decrease to a dose of 137mg/day (half dose) of GOCOVRI for one week, before stopping the medication completely.
  All participants will receive GOCOVRI and they will know that they are on study drug. No placebo group.
Arm/Group | GOCOVRI Half Dose (Week 0-2) | GOCOVRI Full Dose (Week 2-4) | GOCOVRI Half Dose (Week 4-5)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 2/8 | 1/6 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GOCOVRI Half Dose (Week 0-2) (N=8) | GOCOVRI Full Dose (Week 2-4) (N=6) | GOCOVRI Half Dose (Week 4-5) (N=5)
Dry mouth (xerostomia) (General disorders) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT04387773/Prot_SAP_000.pdf